CLINICAL TRIAL: NCT07111169
Title: Selective Attention Deficits and Neuromodulation in Major Depressive Disorder: Using EEG and MRI-guided iTBS Study
Brief Title: Neuromodulation and Attention Deficits in MDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Beckerlab, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BAM_lab_MDD_01
Record Dates: First submitted 2025-07-31; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Major Depression Disorder; Cognitive Deficits; Selective Attention
Keywords: iTBS; EEG; MDD
MeSH Terms: conditions — Cognition Disorders | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants did not know whether they were receiving iTBS or sham; Intervention Operator knew whether the participants were receiving iTBS or sham; and Outcomes Assessor who evaluated HAMD/HAMA and analyzed the scale data did not know which group each MDD participant was assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MDD subjects in the active group undergo 10 days of MRI-guided iTBS intervention (Experimental): Neuronavigation procedure: During the iTBS treatment, the high-resolution T1-weighted scans of each subject will be uploaded to the BrainSight neuronavigation system (version 2.4.11), adjusted, and remodelled into a three-dimensional model. Then, the neuronavigation system is calibrated and validated on the subject. Next, we localized each participant's left-lateral dlPFC stimulation target using Talairach coordinates (-45, 45, 35). The head position is standardized using the nasal tip, sinuses, and bilateral ear screens as baseline markers, and the location of the target on the scalp is identified in each participant's natural space anatomical image. In the end, we observe on the computer screen whether the coil position is placed above the target through the navigation software and artificially control the coil to be tangent to the skull, with the center of the figure-of-eight coil always directly above the target.
  Interventions: Device: intermittent theta burst stimulation (iTBS) intervention
- MDD controls in the sham-iTBS group receive the same intervention but Beam F3 site. (Sham Comparator): Target Localization and Cap Placement Procedure: The stimulation target was the EEG 10-20 coordinate F3, corresponding to the probabilistic location of the left dorsolateral prefrontal cortex (DLPFC). We localized this site using the Beam F3 method and a TMS elastic cap (patent no. 201120150878.5, Wuhan YIRUIDE Medical Equipment Co., Ltd.), and verified it with the F3 electrode on the standard EEG cap. Before the first session, the elastic cap was aligned using anatomical landmarks (nasion, inion, and ears), and the F3 position was marked for consistent coil placement. This standardized approach ensured precise and repeatable targeting across TMS sessions.
  Interventions: Device: intermittent theta burst stimulation (iTBS) intervention

INTERVENTIONS:
Device: intermittent theta burst stimulation (iTBS) intervention — iTBS protocol: Intervention with an 80-120% resting threshold was used. In the active group, the left dlPFC was selected as the stimulation site and a stimulation protocol with iTBS parameters was given. This was a neuro-modulation protocol of excitatory sequences, with theta burst stimulation at 50 Hz, repeated at 5 Hz, stimulation for 2 s with an interval of 8 s, for a total of 1,800 pulses, with a treatment time of about 20 min/session, two sessions per day, with a15-30 min rest between sessions, and five consecutive days of treatment per week, with a rest of 2 days, and two weeks of treatment.

SUMMARY:
Multimodal study (Behavior, TMS, EEG) combining a sham-controlled intermittent theta burst stimulation (iTBS) intervention with an additional-singleton task and EEG to evaluate whether left dorsolateral prefrontal cortex (DLPFC) stimulation enhances cognitive control and modulates maladaptive attention processes in MDD and whether the effects are influenced by neuronavigated versus manual (Beam F3 method) localization of the stimulation site.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is associated with impaired selective attention and disrupted top-down control, yet the underlying neurophysiological mechanisms remain poorly understood. The present double-blind, sham-controlled trial will test whether iTBS over the left DLPFC, an FDA-approved rTMS site, can restore top-down distractor suppression in MDD (active-iTBS: n = 30; sham-iTBS: n = 30). Neuronavigated iTBS will be delivered across sessions, and effects will be assessed on the behavioral level (additional singleton paradigm) and the neurophysiological level (using concomitant EEG). Key aim of the project is to compare neuronavigated (active-iTBS) versus manual (Beam F3 method, sham-iTBS group) localization of the stimulation site.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years
* Right-handed
* Normal or corrected normal visual acuity
* MDD: meet the proposed DSM-5 MDD criteria, unmedicated or stable medicated within the last one month. Healthy subjects without any past or present psychiatric or neurological disorders.

Exclusion Criteria:

* Diagnosis of other severe mental disorders, such as schizophrenia, bipolar disorder, neurodevelopmental disorder, etc.
* high suicidal risk
* Unnormal intellectual functioning, auditory impairments,
* Have received neuromodulation, such as Modified Electroconvulsive Therapy (MECT), or any psychotherapy within the past 6 months.
* Only for the active-iTBS group: have a contraindication to MRI scanning (e.g., metal implants, claustrophobia or other conditions that make them inappropriate for MRI scanning).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Depression severity following two weeks of iTBS treatment. | 60-90 minutes before the first iTBS treatment and 60-90 minutes after last iTBS treatment.
  Depression severity will be assessed, using 24-item Hamilton Depression Scale (HAMD-24) before and after the iTBS intervention. Changes will be computed as (pre-treatment score - post-treatment score)/pre-treatment score × 100%). We hypothesize that the neuronaviogated group has a better treatment effect indexed by the mean HAMD subtraction rate than the sham-control group.

SECONDARY OUTCOMES:
Intervention-related ERPs changes in the additional singleton task after 2 weeks of active/sham iTBS treatment. | 30-60 minutes before the first iTBS treatment and 30-60 minutes after last iTBS treatment.
  Neuromodulation-induced iTBS changes will be measured by the probability cueing effects in the additional singleton task with ERP effects. N2pc and Pd components will be used to quantify attentional selection and distractor suppression. These ERP components reflect the neural mechanisms of spatial attention in MDD.
Intervention-related brain connectivity after 2 weeks of active/sham iTBS treatment. | 30-60 minutes before the first iTBS treatment and 30-60 minutes after last iTBS treatment.
  During the additional singleton task, we will measure network-level connectivity patterns between attention-related brain regions (e.g., fronto-parietal and sensory integration systems). Directed or undirected EEG connectivity methods (e.g., phase synchronization, Granger causality, or sPDC) will be applied to assess iTBS-induced changes in intrinsic attentional network architecture in MDD.
Intervention-related behavior changes in the additional singleton task after 2 weeks of active/sham iTBS treatment. | 30-60 minutes before the first iTBS treatment and 30-60 minutes after the last iTBS treatment.
  Neuromodulation-induced iTBS changes will also be measured in RTs. We aim to examine whether the different RT effects in both groups occur between the pre-iTBS and post-iTBS conditions. For the between-group effect, compared to the sham-iTBS group, the active-iTBS group has faster RTs and statistical learning effects (e.g., subtraction RTs from the low-minus-high-probability distractor locations).

CONTACTS AND LOCATIONS:
Locations (1):
- The Clinical Hospital of Chengdu Brain Science Institute, Chengdu Fourth People's Hospital, Jiujiang Branch (Chengdu Mental Health Center), Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided